CLINICAL TRIAL: NCT00001302
Title: A Phase I Study of Infusional Chemotherapy With the P-Glycoprotein Antagonist PSC 833
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 920268; 92-C-0268
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-06

CONDITIONS: Breast Cancer; Kidney Neoplasm; Lymphoma; Neoplasm Metastasis; Ovarian Cancer
Keywords: Vinblastine; Multidrug Resistance; Resistance Reversal; Pgp Blocker; Pharmacokinetics; Cyclosporine; Drug Interactions
MeSH Terms: conditions — Breast Neoplasms; Kidney Neoplasms; Lymphoma; Neoplasm Metastasis; Ovarian Neoplasms | interventions — valspodar

INTERVENTIONS:
Drug: PSC 833

SUMMARY:
The clinical study entitled "A Phase I Study of Infusional Chemotherapy with the P-glycoprotein Antagonist PSC 833" seeks to determine the maximum tolerated dose for a proposed P-glycoprotein antagonist, PSC 833. PSC 833 is a cyclosporine analogue which is purportedly non-nephrotoxic and non-immunosuppressive. It has been shown in in-vitro studies to enhance chemosensitivity as well as cyclosporine and to be far better at increasing intracellular drug accumulation than the concentrations of verapamil which are clinically achievable. The purpose of this study is to define the maximum tolerated dose in combination with vinblastine, and to determine how the drug affects the pharmacokinetics of vinblastine. PSC 833 will most likely reduce the clearance of vinblastine, as reported for the parent compound, cyclosporine. This effect will increase the area under the curve (AUC) of vinblastine, may increase toxicity, and requires that the escalation scheme for PSC 833 be a conservative one. Initially, a 120 hour infusion of vinblastine will be given alone. Then 8 days of PSC 833 will follow to allow monitoring of adverse effects of PSC 833 alone. This first cycle of vinblastine will be given in the absence of PSC 833; in second and subsequent cycles both agents will be combined. Escalation of the PSC 833 will continue until a target concentration is reached, or until the maximum tolerated dose is reached. Clinical responses will be monitored in order to provide the best possible medical care to our patients.

DETAILED DESCRIPTION:
The clinical study entitled "A Phase I Study of Infusional Chemotherapy with the P-glycoprotein Antagonist PSC 833" seeks to determine the maximum tolerated dose for a proposed P-glycoprotein antagonist, PSC 833. PSC 833 is a cyclosporine analogue which is purportedly non-nephrotoxic and non-immunosuppressive. It has been shown in in vitro studies to enhance chemosensitivity as well as cyclosporine and to be far better at increasing intracellular drug accumulation than the concentrations of verapamil which are clinically achievable. The purpose of this study is to define the maximum tolerated dose in combination with vinblastine, and to determine how the drug affects the pharmacokinetics of vinblastine. PSC 833 will most likely reduce the clearance of vinblastine, as reported for the parent compound, cyclosporine. This effect will increase the area under the curve (AUC) of vinblastine, may increase toxicity, and requires that the escalation scheme for PSC 833 be a conservative one. Initially, a 120 hour infusion of vinblastine will be given alone. Then 8 days of PSC 833 will follow to allow monitoring of adverse effects of PSC 833 alone. This first cycle of vinblastine will be given in the absence of PSC 833; in second and subsequent cycles both agents will be combined. Escalation of the PSC 833 will continue until a target concentration is reached, or until the maximum tolerated dose is reached. Clinical responses will be monitored in order to provide the best possible medical care to our patients.

ELIGIBILITY:
Biopsy proven metastatic cancer, for whom no better therapy exists. All patients are eligible. Enrollment of patients with kidney, breast, ovarian cancers, and lymphomas is encouraged.

A life expectancy of at least 16 weeks, and a performance status (Karnofsky scale) of 70% or greater. Patients without rapidly growing disease.

Any prior therapy except for previous bone marrow transplantation.

WBC greater than 3,000/mm3 and ACG greater than 1,000/mm3; platelets greater than 100,000/mm3.

Creatinine Clearance greater than 50 ml/min; bilirubin less than 1.5 mg/dl; SGOT less than 70u/L; SGPT less than 80u/L.

A signed informed consent and geographic accessibility for the patient to return for follow up and treatment.

No history of brain metastases.

Not currently receiving treatment with the following agents or any other agent known to significantly interact with cyclosporine, and treatment cannot be discontinued, or changed to another therapeutically equivalent allowable drug: acetazolamide, barbiturates, corticosteroids, diltiazem, erythromycin, fluconazole, ketoconazole, nicardipine, phenothiazines, phenytoin, rifampin, sulfonamides, trimethoprim, verapamil, tamoxifen, progesterone, quinine, quinidine, or amiodarone.

No symptomatic peripheral neuropathy (grade 2 or greater arising from prior vinca alkaloid therapy).

No positive serology for HIV.

No ongoing pregnancy or unwillingness to practice adequate contraception.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80
Dates: Start 1992-09; Study Completion 2002-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Yahanda AM, Alder KM, Fisher GA, Brophy NA, Halsey J, Hardy RI, Gosland MP, Lum BL, Sikic BI. Phase I trial of etoposide with cyclosporine as a modulator of multidrug resistance. J Clin Oncol. 1992 Oct;10(10):1624-34. doi: 10.1200/JCO.1992.10.10.1624. PMID 1403040
- [Background] Samuels BL, Mick R, Vogelzang NJ, Williams SF, Schilsky RL, Safa AR, O'Brien SM, Ratain MJ. Modulation of vinblastine resistance with cyclosporine: a phase I study. Clin Pharmacol Ther. 1993 Oct;54(4):421-9. doi: 10.1038/clpt.1993.169. PMID 8222485
- [Background] Piwnica-Worms D, Chiu ML, Budding M, Kronauge JF, Kramer RA, Croop JM. Functional imaging of multidrug-resistant P-glycoprotein with an organotechnetium complex. Cancer Res. 1993 Mar 1;53(5):977-84. PMID 8094997